CLINICAL TRIAL: NCT06047444
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Multicenter, Parallel-group Study With Extension Phase to Evaluate the Efficacy and Safety of Dysport® for the Prevention of Chronic Migraine in Adult Participants
Brief Title: A Study to Evaluate the Effectiveness and Safety of Dysport® for the Prevention of Chronic Migraine in Adults
Acronym: C-BEOND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CLIN-52120-463; 2023-504827-17-00 (EU CTIS Number)
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Migraine
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dysport® dose "A" (Experimental): Participant will receive four treatment cycles, each separated by an interval of 12 weeks.
  Double-blind placebo-controlled (DBPC) Phase: Dysport® dose "A" administered intramuscularly on Day 1 and Week 12.
  Extension Phase: Dysport® dose "A" administered intramuscularly at Week 24 and Week 36 (final follow-up at Week 48)
  Interventions: Biological: Botulinum toxin type A
- Dysport® dose "B" (Experimental): Participant will receive four treatment cycles, each separated by an interval of 12 weeks.
  DBPC Phase: Dysport® dose "B" administered intramuscularly on Day 1 and Week 12.
  Extension Phase: Dysport® dose "B" administered intramuscularly at Week 24 and Week 36 (final follow-up at Week 48)
  Interventions: Biological: Botulinum toxin type A
- Placebo - Dysport dose "A" (Placebo Comparator): Participant will receive four treatment cycles, each separated by an interval of 12 weeks.
  DBPC Phase: Placebo dose "A" administered intramuscularly on Day 1 and Week 12
  Extension Phase: Dysport® dose "A" administered intramuscularly at Week 24 and Week 36 (final follow-up at Week 48)
  Interventions: Other: Placebo; Biological: Botulinum toxin type A
- Placebo - Dysport dose "B" (Placebo Comparator): Participant will receive four treatment cycles, each separated by an interval of 12 weeks.
  DBPC Phase: Placebo dose "B" administered intramuscularly on Day 1 and Week 12.
  Extension Phase: Dysport® dose "B" administered intramuscularly at Week 24 and Week 36 (final follow-up at Week 48).
  Interventions: Other: Placebo; Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — Dose "A" Unit/Injection (U/I), Intramuscular (IM) on every 12 weeks during a period of 36 weeks with a total of 4 injections.
  Other Names: Dysport®
  Arms: Dysport® dose "A"
Biological: Botulinum toxin type A — Dose "B" U/I, IM on every 12 weeks during a period of 36 weeks with a total of 4 injections.
  Other Names: Dysport®
  Arms: Dysport® dose "B"
Other: Placebo — "0" U/I, IM on Day 1 and Week 12 with a total of 2 injections.
  Arms: Placebo - Dysport dose "A"; Placebo - Dysport dose "B"
Biological: Botulinum toxin type A — Dose "A" U/I, IM at Week 24 and Week 36 with a total of 2 injections.
  Other Names: Dysport®
  Arms: Placebo - Dysport dose "A"
Biological: Botulinum toxin type A — Dose "B" U/I, IM at Week 24 and Week 36 with a total of 2 injections.
  Other Names: Dysport®
  Arms: Placebo - Dysport dose "B"

SUMMARY:
The purpose of this study is to understand the safety and effectiveness of the study drug, Dysport® when compared with placebo in preventing chronic migraine.

A migraine is a headache with severe throbbing pain or a pulsating sensation, usually on one side of the head, and is often accompanied by feeling or being sick and a sensitivity to bright lights and sound.

Chronic migraine is defined as having at least 15 days of headache a month with at least 8 of those days being migraine headache days.

Migraines are caused by a series of events which cause the brain to get stimulated/activated, which results in the release of chemicals that cause pain. Dysport® is a formulation of Botulinum toxin type A (BoNT-A), a medication that stops the release of these chemical messengers.

The study will consist of 3 periods:

1. A 'screening period' of 6 to 12 weeks to assess whether the participant can take part to the study and requires 1 visit.
2. A first Treatment Phase of 24 weeks. On Day 1 and at Week 12 of the first Treatment Phase, participants will receive injections into various muscles across the head, neck, face and shoulders.

   The injections will contain either a dose "A" or dose "B" of Dysport® or a placebo (an inactive substance or treatment that looks the same as, and is given in the same way as, an active drug or intervention/treatment being studied). Participants will make 4 visits to the clinic in person and have 4 remote (online) visits.
3. A second Treatment Phase of 24 weeks (extension phase). At Week 24 and at Week 36, all participants will get Dysport® (dose "A" or dose "B").

There will be 3 in person visits and 4 remote visits.

Participants will need to complete an e-diary and questionnaires throughout the study. Participants will undergo blood samplings, urine collections, physical examinations, and clinical evaluations.

They may continue some other medications, but the details need to be recorded. The total study duration for a participant will be up to 60 weeks (approx. 14 months).

ELIGIBILITY:
Inclusion Criteria :

* Participant must be ≥18 years of age inclusive, at the time of signing the informed consent and privacy/data protection documentation
* Participant has a diagnosis for more than 12 months, prior to screening visit, of chronic migraine according to the International Classification of Headache Disorders definition and diagnostic criteria
* Migraine onset occurred when participant was <50 years of age
* Has baseline number of monthly headache days (MHD) ≥15 and baseline number of monthly migraine days (MMD) of ≥8, using eDiary data collected during the 4 weeks nearest to randomisation on Day 1 (but prior to randomisation)
* Has baseline number of valid diary days ≥22 days collected during the 4 weeks nearest to randomisation on Day 1
* Participant must have previously used, or is currently using, preventive treatment for migraine (pharmacological) (i.e. non-naïve) prior to start of screening eDiary

Exclusion Criteria :

* History or current diagnosis of migraine with brainstem aura, retinal migraine, complications of migraine, tension-type headache, trigeminal autonomic cephalalgias, hypnic headache, hemicrania continua, or new daily persistent headache
* Headache attributed to another disorder (e.g. secondary headaches), except medication overuse headache, which is permitted
* Use of any of the following medications in the specified timeframe prior to start of the screening daily headache eDiary:

Within 24 weeks

* i. Botulinum toxin for migraine (or for any other medical/aesthetic reason within 16 weeks)

Within 12 weeks

* i. CGRP antagonists (monoclonal antibody or gepant) for preventive treatment of migraine (acute treatment of headache/migraine with a gepant is permitted but limited to no more than 6 days per month (i.e 6 days per each 4-week period with gepant intake))
* ii. Cannabidiol or other types of cannabinoids

Within 4 weeks

* i. Anaesthetic or steroid injection in any region targeted for injection with study intervention
* ii. Use of medical device to treat migraine (e.g. non-invasive neuromodulation therapies such as nerve stimulation (gammaCore), transcranial magnetic stimulation (cephaly), external trigeminal nerve stimulation, transcutaneous electrical nerve stimulation, and peripheral neuroelectrical stimulation)
* iii. Other interventions for migraine assessed to interfere with study evaluations (e.g. acupuncture in head and neck region, cranial traction, nociceptive trigeminal inhibition, occipital nerve block treatments, and dental splints for headache)
* iv. Use of opioids or barbiturates for more than 2 days/month. Note: participants are permitted to take one concomitant migraine preventative treatment (not listed above); however, the dose of this medication should be stable for ≥3 months before start of the screening eDiary
* Known history of treatment failure to more than four medications prescribed for the prevention of migraine (two of which have different mechanisms of action) or known history of treatment failure to botulinum toxin prescribed for the prevention of migraine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline at week 24 in monthly migraine days (MMD) | Every 4 weeks from Week 4 (Weeks 1-4) to Week 24 (Weeks 21-24)
  The monthly migraine days (MMD) is assessed by eDiary, completed every day by the participant, to evaluate the efficacy of Dysport® compared to placebo.

SECONDARY OUTCOMES:
Change from baseline in MMD of ≥50% | Every 4 weeks from Week 4 (Weeks 1-4) to Week 24 (Weeks 21-24)
  The monthly migraine days (MMD) is assessed by a daily eDiary.
Change from baseline in MMD of ≥75% | Every 4 weeks from Week 4 (Weeks 1-4) to Week 24 (Weeks 21-24)
  The monthly migraine days (MMD) is assessed by a daily eDiary.
Cumulative number of MMD | From Day 1 to Week 24
  The cumulative number of monthly migraine days (MMD) is assessed by a daily eDiary.
Change from baseline in MMD of moderate or severe intensity | Every 4 weeks from Week 4 (Weeks 1-4) to Week 24 (Weeks 21-24)
  The intensity of MMD is assessed by a daily eDiary.
Change from baseline in the number of MMD over the last 12 weeks prior to Week 24 | From Week 13 - 24
  The monthly migraine days (MMD) is assessed by a daily eDiary.
Change from baseline in monthly headache days (MHD) of moderate or severe intensity | Every 4 weeks from Week 4 (Weeks 1-4) to Week 24 (Weeks 21-24)
  The intensity of monthly headache days (MHD) is assessed by a daily eDiary.
Change from baseline in MHD of moderate or severe intensity of ≥50% | Every 4 weeks from Week 4 (Weeks 1-4) to Week 24 (Weeks 21-24)
  The intensity of monthly headache days (MHD) is assessed by a daily eDiary.
Change from baseline in MHD of moderate or severe intensity of ≥75% | Every 4 weeks from Week 4 (Weeks 1-4) to Week 24 (Weeks 21-24)
  The intensity of monthly headache days (MHD) is assessed by a daily eDiary.
Cumulative number of MHD of moderate or severe intensity | From Day 1 to Week 24
  The cumulative number of monthly headache days (MHD) is assessed by a daily eDiary.
Change from baseline in the number of days per month of acute migraine medication intake | Every 4 weeks from Week 4 (Weeks 1-4) to Week 24 (Weeks 21-24)
  The acute migraine specific medication intake will be recorded in the daily eDiary. Acute migraine medication is defined as triptan, ergotamine, gepant, or ditan.
Headache medication overuser (yes, no) | Every 4 weeks from Week 4 (Weeks 1-4) to Week 24 (Weeks 21-24)
  The headache medication overuse will be assessed by a concomitant medication log completed at each visit and acute medication taken to treat acute attack will be recorded in the daily eDiary. The headache medication overuse is defined as a participant with ≥10 days/month if ergotamine, triptan, gepant, ditan, opioid or combination analgesic, or ≥15 days/month if non-opioid analgesic (such as paracetamol, aspirin, NSAID)
Use of acute migraine medication (yes or no) | Every 4 weeks from Week 4 (Weeks 1-4) to Week 24 (Weeks 21-24)
  The use of acute migraine medication will be recorded in the daily eDiary.
Patient's Global Impression of Change (PGIC) score | At Weeek 12 and Week 24
  The PGIC will be assessed by a questionnaire (7-point scale, score of 1 indicates very much improved and score of 7 indicates very much worse)
Change from baseline of ≥1 and ≥2 grades in PGIC score | At Weeek 12 and Week 24
  The PGIC will be assessed by a questionnaire (7-point scale, score of 1 indicates very much improved and score of 7 indicates very much worse)
Change from baseline in role function restrictive (RFR) domain of Migraine Specific Quality of Life (MSQ) Questionnaire | At Weeek 12 and Week 24
  The MSQ will be assessed by a questionnaire (Scores range from 0-100, higher scores indicate a better quality of life)
Change from baseline in role function-preventive (RFP) domain of MSQ Questionnaire | At Week 12 and Week 24
  The MSQ will be assessed by a questionnaire (Scores range from 0-100, higher scores indicate a better quality of life)
Change from baseline in emotional function (EF) domain of MSQ Questionnaire | At Week 12 and Week 24
  The MSQ will be assessed by a questionnaire (Scores range from 0-100, higher scores indicate a better quality of life)
Change from baseline in total MSQ score | At Weeek 12 and Week 24
  The MSQ will be assessed by a questionnaire (Scores range from 0-100, higher scores indicate a better quality of life)
Change in MSQ score to the minimally important change (MIC) thresholds | At Weeek 12 and Week 24
  The MSQ will be assessed by a questionnaire (Scores range from 0-100, higher scores indicate a better quality of life)
Change from baseline in total 6-item Headache Impact Test (HIT-6) score | At Week 12 and Week 24
  The HIT-6 will be assessed by a questionnaire (scores range from 36-78 and higher scores indicate a greater impact of headache on subject's life)
Change from baseline in HIT-6 score to MIC thresholds | At Weeek 12 and Week 24
  The HIT-6 will be assessed by a questionnaire (scores range from 36-78 and higher scores indicate a greater impact of headache on subject's life)
Change from baseline in Short Form 12 (SF-12) Questionnaire score | At Weeek 12 and Week 24
  The SF-12 will be assessed by a questionnaire (scores range from 0-100, with higher scores indicating better functioning)
Chronic migraine status | At Week 24 (Week 21-24)
  Chronic migraine status will be assessed by the daily eDiary and defined as number of participants with ≥15 MHD and ≥8 MMD
Time to onset of effect | From first time point post randomisation to Week 24
  Time to onset of effect is defined as the first time point post randomisation where MMD is reduced from baseline ≥50%
Incidence of Treatment emergent adverse event (TEAEs) | Up to Week 24
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of Participants with clinically significant changes in vital signs | From baseline up to Week 24
  Percentage of participants with clinically significant changes in vital signs will be reported. The clinical significance will be graded by the investigator.
Percentage of participants with clinically significant laboratory parameters (blood chemistry, haematology) | From baseline up to Week 24
  Percentage of participants with clinically significant change in laboratory parameters (blood chemistry, hematology and coagulation) will be reported. The clinical significance will graded by the investigator.
Treatment-emergence of suicidal ideation/suicidal behaviour | From baseline up to Week 24
  It will be assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) questionnaire that consists of 4 subscales:
  1. Ideation severity subscale: questions answered yes/no, severity of ideation scored 1-5 with 5 being most severe
  2. Intensity of ideation subscale : scores range from 2-25 with higher scores indicating more severe intensity of ideation.
  3. Suicide behaviour subscale:4 types of suicidal behaviours are scored yes/no
  4. Behaviour Lethality subscale: actual lethality/medical damage scores 0-5, with 5 being most severe ( death) and potential lethality scores 0-2 with 2 being more potentially lethal.
Percentage of participants with binding antibodies to Dysport® | At Week 24
  Presence of binding antibodies will be assessed using a validated method of electrochemiluminescence assay (ECLA).
Percentage of participants with neutralising antibodies to Dysport® | At Week 24
  It will be performed only for confirmed positive samples with ECLA (confirmation of the presence of binding antibodies). Presence of neutralizing antibodies will be assessed using a validated cell-based assay (CBA).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (120):
- United States (72):
  - Central Research Associates, Birmingham, Alabama
  - CCT Research, Phoenix, Arizona
  - HonorHealth Neurology, Scottsdale, Arizona
  - Hope Clinical Research, LLC, Canoga Park, California
  - Axiom Research LLC, Colton, California
  - Fullerton Neurological Center, Fullerton, California
  - Neurology Center of North Orange County, Fullerton, California
  - The Los Angeles Headache Center, Los Angeles, California
  - SDS Clinical Trials, Orange, California
  - 840011, Palo Alto, California
  - Stanford University School of Medicine - Stanford Cardiovascular Institute (CVI), Palo Alto, California
  - Alliance Clinical San Diego (Acclaim Clinical Research), San Diego, California
  - University of Colorado Hospital - Neurology Clinic, Aurora, Colorado
  - Yale University School of Medicine, East Hartford, Connecticut
  - Hasbani Neurology, New Haven, Connecticut
  - New England Institute for Neurology and Headache (NEINH)/Medical Practice, Stamford, Connecticut
  - Visionary Investigators Network (VIN), Aventura, Florida
  - Velocity Clinical Research - Hallandale Beach, Hallandale, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Neurology Clinical Research, Inc., Hollywood, Florida
  - Clinical Neuroscience Solutions Healthcare, Inc (CNS Healthcare, INC), Jacksonville, Florida
  - University of Miami Leonard M. Miller School of Medicine - Professional Arts Center, Miami, Florida
  - Quantum Clinical Trials, Miami Beach, Florida
  - Clinical Neuroscience Solutions, Inc ((CNS Healthcare) - Psychiatry), Orlando, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - USF Health-Morsani Center, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Headache Wellness Center, Greensboro, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Chicago Headache Center & Research, Chicago, Illinois
  - Robbins Headache Clinic, Riverwoods, Illinois
  - MD Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Comprehensive Neurology Services, Frederick, Maryland
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center - Arnold Pain Management, Brookline, Massachusetts
  - Neurology Center of NE,PC - Neurology, Foxborough, Massachusetts
  - Mass Institute of Clinical Research, Westborough, Massachusetts
  - New England Regional Headache Center, Inc., Worcester, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Minneapolis Clinic of Neurology, Burnsville, Minnesota
  - Papillion Research Center, Papillion, Nebraska
  - WR-CRCN, Las Vegas, Nevada
  - Alliance Clinical Las Vegas (Excel Clinical Research), Las Vegas, Nevada
  - Dent Neurosciences Research Center, Inc., Amherst, New York
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Nuvance Health Medical Practice, Poughkeepsie, New York
  - Rochester Clinical Research, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Blue Sky MD, Hendersonville, North Carolina
  - Headache Center of Hope, Cincinnati, Ohio
  - OrthoNeuro, New Albany, Ohio
  - Helios Clinical Research, Wooster, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Thomas Jefferson University Hospital - Jefferson Hospital for Neuroscience - Jefferson Neurology Associates - Neurology, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center - North Charleston, North Charleston, South Carolina
  - Neurology Clinic, PC, Cordova, Tennessee
  - KCA Neurology, PLLC, Franklin, Tennessee
  - Helios Clinical Research LLC (Helios CR, Inc. Jackson TN), Jackson, Tennessee
  - Herzog, Steven MD, Dallas, Texas
  - Texas Neurology, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Lone Star Neurology, Frisco, Texas
  - Clinical Trial Network, Houston, Texas
  - Research Your Health, Plano, Texas
  - J. Lewis Research Inc.-Foothill, Salt Lake City, Utah
  - Metrodora Institute, West Valley City, Utah
  - Inova Medical Group - Neurology, Fairfax, Virginia
  - MedStar Health - Department of Neurology, Columbia, Washington
  - Frontier Clinical Research, LLC, Kingwood, West Virginia
  - BCN Research, LLC, Greenfield, Wisconsin
  - Neuroscience Group of Northeast Wisconsin-Neenah, Neenah, Wisconsin
- Canada (5):
  - Centricity Research Halifax Multispecialty, Halifax
  - Genge Partners Inc., Montreal
  - CARe Clinic-Calgary, Red Deer
  - Bluewater Clinical Research Group Inc., Sarnia
  - Royal Julilee Hospital, Victoria
- Czechia (9):
  - Neurologie Brno s.r.o., Brno
  - Pratia Brno s.r.o., Brno
  - NeuropsychiatrieHK, s.r.o., Hradec Králové
  - Nemocnice Jihlava, p.o., Jihlava
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Axon Clinical, s.r.o., Prague
  - DADO MEDICAL s.r.o., Prague
  - Fakultni Thomayerova nemocnice, Prague
  - Institut neuropsychiatricke pece, Prague
- Georgia (6):
  - Ltd "Health", Batumi
  - ISR-GEO Med Res Clin Healthycore, Tbilisi
  - "Pineo Medical Ecosystem" LTD, Tbilisi
  - LTD New Hospitals, Tbilisi
  - LTD S.Khechinashvili University Hospital, Tbilisi
  - Multprofil Clinic Consilium Medulla, Tbilisi
- Germany (6):
  - Charité - Universitätsmedizin Berlin KöR, Berlin
  - Emovis GmbH, Berlin
  - Universitätsmedizin Greifswald, Greifswald
  - Curiositas ad sanum Studien- und Beratungs GmbH Haag i.OB, Haag in Oberbayern
  - Vitos Orthopaedische Klinik Kassel, Kassel
  - LMU - Klinikum der Universität München - Campus Grosshadern, München
- Italy (6):
  - Ospedale Bellaria, IRCCS Istituto delle Scienze Neurologiche, AUSL di Bologna, Bologna
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli, Napoli
  - IRCCS C.Mondino, Istituto Neurologico Nazionale, Fondazione, Pavia
  - Istituto Neurologico Mediterraneo - NEUROMED, Istituto di Ricovero e Cura a Carattere Scientifico, Pozzilli
  - IRCCS San Raffaele Pisana, Roma
  - PU Campus Bio-Medico di Roma, Roma
- Poland (8):
  - Centrum Medyczne Neuromed Pawel Lisewski, Bydgoszcz
  - Synexus Polska Sp. z o.o., Gdynia
  - Centrum Medyczne Pratia Katowice, Katowice
  - Krakowska Akademia Neurologii Sp. z o.o., Krakow
  - Krakowskie Centrum MedyczneSp.z o.o, Krakow
  - Pratia MCM Krakow, Krakow
  - Indywidualna Praktyka Lekarska dr hab. med. Anna Szczepanska-Szerej, Lublin
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. z o.o. S.K., Oświęcim
- Spain (6):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Regional De Malaga, Málaga
  - Hospital Universitario Virgen De La Macarena, Seville
  - Hospital Clinico Universitario De Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (2):
  - University Hospitals Sussex NHS Foundation Trust - Royal Sussex County Hospital, Brighton
  - King's College Hospital (KCH) NHS Foundation Trust, Brixton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/